CLINICAL TRIAL: NCT01985425
Title: Colchicine For Prevention of Perioperative Atrial Fibrillation in Patients Undergoing Thoracic Surgery Pilot Study.
Acronym: COP-AF Pilot
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COP-AF Pilot
Record Dates: First submitted 2013-11-08; First posted 2013-11-15 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Atrial Fibrillation; Thoracic Surgery
MeSH Terms: conditions — Atrial Fibrillation | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Colchicine (Experimental): On the day of surgery, the intervention group will receive 2 doses of colchicine 0.6 mg orally. The first dose will be administered within 4 hours before surgery. The second dose will be given between 6:00PM and 11:59PM after surgery. All patients will receive colchicine 0.6 mg or placebo twice daily orally for 10 days.
  Interventions: Drug: Colchicine 0.6 mg
- Placebo Colchicine (Placebo Comparator): On the day of surgery, the intervention group will receive 2 doses of colchicine placebo 0.6 mg orally. The first dose will be administered within 4 hours before surgery. The second dose will be given between 6:00PM and 11:59PM after surgery. All patients will receive colchicine 0.6 mg or placebo twice daily orally for 10 days.
  Interventions: Drug: Placebo Colchicine

INTERVENTIONS:
Drug: Colchicine 0.6 mg
  Other Names: Brand names: PMS Colchicine, Colchicine TAB 0.6 mg
  Arms: Active Colchicine
Drug: Placebo Colchicine
  Arms: Placebo Colchicine

SUMMARY:
The purpose of this pilot study is to determine the feasibility of comparing colchicine to placebo for the prevention of new onset atrial fibrillation in patients undergoing general thoracic surgery and establish the foundation for a large, multi-centre, clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥55 years of age undergoing intra-thoracic surgery for a resection of tumor in lung.

Exclusion Criteria:

* In AF prior to surgery*,
* Undergoing minor thoracic interventions/ procedures (i.e., chest tube insertion, needle pleural/lung biopsies, or minor chest-wall surgeries), or
* With contraindications to colchicine (i.e., allergy, or myelodysplastic disorders or estimated glomerular filtration rate [e-GFR] <30 mL/min/1.73m)

  * Clarification: Patients with history of AF who are in sinus rhythm during enrollment will be eligible for recruitment. Patients who have no history of AF and are found to be in AF at the time of enrollment will not be eligible.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PJ Devereaux, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - University of Manitoba Health Sciences Centre, Winnipeg, Manitoba
  - St. Joseph Healthcare, St. Joseph Hospital, Hamilton, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Colchicine: On the day of surgery, the intervention group will receive 2 doses of colchicine 0.6 mg orally. The first dose will be administered within 4 hours before surgery. The second dose will be given between 6:00PM and 11:59PM after surgery. All patients will receive colchicine 0.6 mg or placebo twice daily orally for 10 days.
  Colchicine
- Placebo Colchicine: On the day of surgery, the intervention group will receive 2 doses of colchicine placebo 0.6 mg orally. The first dose will be administered within 4 hours before surgery. The second dose will be given between 6:00PM and 11:59PM after surgery. All patients will receive colchicine 0.6 mg or placebo twice daily orally for 10 days.
  Colchicine Placebo
Period: Overall Study
Arm/Group | Active Colchicine | Placebo Colchicine
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Colchicine | Placebo Colchicine | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.89 (7.5) | 68.28 (7.4) | 68.57 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 22 | 55
  Male | 16 | 29 | 45
Region of Enrollment [Number; unit: participants]
  Canada | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Atrial Fibrillation
Description: New atrial fibrillation that results in angina, congestive heart failure, symptomatic hypotension, or that requires treatment with a rate controlling drug, antiarrhythmic drug, or electrical cardioversion, or that lasts for longer than 30 seconds.
Time Frame: Post-operative Day 1 until Postoperative Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Active Colchicine | Placebo Colchicine
Number analyzed (Participants) | 49 | 51
Participants | 5 | 6

2. Secondary Outcome: Death
Time Frame: Post-operative Day 1 until Postoperative Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Active Colchicine | Placebo Colchicine
Number analyzed (Participants) | 49 | 51
Participants | 0 | 0

3. Secondary Outcome: New Onset Atrial Flutter
Description: Replacement of the consistent P waves on 12-lead ECG, or documented telemetry tracing, by saw-tooth flutter waves.
Time Frame: Post-operative Day 1 until Postoperative Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Active Colchicine | Placebo Colchicine
Number analyzed (Participants) | 49 | 51
Participants | 0 | 1

4. Secondary Outcome: Myocardial Injury After Non-Cardiac Surgery (MINS)
Description: Requires one of the following criteria:
  A) Elevated troponin or CK-MB measurement with one or more of the following defining features:
  1. Ischemic signs or symptoms (i.e., chest, arm, neck, or jaw discomfort; shortness of breath, pulmonary edema);
  2. Development of pathologic Q waves present in any two contiguous leads that are >30 milliseconds;
  3. Electrocardiogram (ECG) changes indicative of ischemia (i.e., ST segment elevation [>2 mm in leads V1, V2, or V3 OR >1 mm in the other leads], ST segment depression [>1 mm], OR symmetric inversion of T waves >1 mm) in at least two contiguous leads;
  4. New LBBB; or v. new or presumed new cardiac wall motion abnormality on echocardiography or new or presumed new fixed defect on radionuclide imaging;
  B) Elevated troponin measurement after surgery with no alternative explanation (e.g., pulmonary embolism, sepsis) to myocardial injury
Time Frame: Post-operative Day 1 until Postoperative Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Active Colchicine | Placebo Colchicine
Number analyzed (Participants) | 49 | 51
Participants | 10 | 12

5. Secondary Outcome: Stroke
Description: New focal neurological deficit thought to be vascular in origin with signs and symptoms lasting more than 24 hours and cerebral imaging consistent with acute stroke.
Time Frame: Post-operative Day 1 until Postoperative Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Active Colchicine | Placebo Colchicine
Number analyzed (Participants) | 49 | 51
Participants | 0 | 0

6. Secondary Outcome: Transient Ischemic Attack (TIA)
Description: New focal neurological deficit thought to be vascular in origin with signs and symptoms lasting less than 24 hours.
Time Frame: Post-operative Day 1 until Postoperative Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Active Colchicine | Placebo Colchicine
Number analyzed (Participants) | 49 | 51
Participants | 0 | 0

7. Secondary Outcome: Post-operative Infection
Time Frame: Post-operative Day 1 until Postoperative Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Active Colchicine | Placebo Colchicine
Number analyzed (Participants) | 49 | 51
Participants | 6 | 8

ADVERSE EVENTS:
Arm/Group | Active Colchicine | Placebo Colchicine
Serious Adverse Events (participants affected / at risk) | 3/49 | 3/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Colchicine (N=49) | Placebo Colchicine (N=51)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
fall (Nervous system disorders) | 2 (2) | 0 (0)
unconsciousness (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes